CLINICAL TRIAL: NCT00049101
Title: A Phase I/II Study Of OSI-774 In Combination With Oxaliplatin, And 5-Fluourouracil In Patients With Metastatic Colorectal Carcinoma
Brief Title: Erlotinib and Combination Chemotherapy in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000257808; MSKCC-02039; NCI-5371
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Erlotinib Hydrochloride; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: erlotinib hydrochloride
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Combining erlotinib with combination chemotherapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining erlotinib with oxaliplatin, leucovorin, and fluorouracil in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of erlotinib when administered with oxaliplatin, leucovorin calcium, and fluorouracil in patients with metastatic colorectal cancer.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine any antitumor activity of this regimen in these patients.
* Determine the time to progression in patients treated with this regimen.
* Determine the objective response rate and response duration in patients treated with this regimen.
* Determine the safety and tolerability of this regimen in these patients.

OUTLINE: This is a dose-escalation study of erlotinib.

* Phase I: During the first week of the first course only, patients receive oral erlotinib daily alone. Patients then begin the regular schedule comprising oral erlotinib daily, oxaliplatin IV over 2 hours on day 1, and leucovorin calcium IV over 2 hours and fluorouracil IV over 22 hours on days 1 and 2. Treatment repeats every 2 weeks for at least 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive erlotinib at the MTD plus oxaliplatin, leucovorin calcium, and fluorouracil as in phase I. Erlotinib may be administered alone if toxicity is caused by oxaliplatin, leucovorin calcium, and fluorouracil.

Patients are followed for at least 6 months or until disease progression.

PROJECTED ACCRUAL: A total of 4-18 patients will be accrued for phase I of this study within 1-4 months. A total of 50 patients will be accrued for phase II of this study within 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colon or rectal cancer

  * Metastatic or unresectable disease
* Unidimensionally measurable disease required for phase II only

  * At least 20 mm by x-ray, CT scan, MRI, or photography
  * The following are not considered measurable:

    * Pleural effusion or ascites
    * Osteoblastic lesions
    * Evidence of disease on bone scan alone
    * Progressive irradiated lesions alone
    * Bone marrow involvement
    * Brain metastases
    * Malignant hepatomegaly by physical exam alone
    * Chemical markers (e.g., carcinoembryonic antigen)
  * Recurrent disease after surgery or radiotherapy is considered measurable as long as the following criteria are met:

    * At least 4 weeks since prior surgery or radiotherapy
    * Measurable disease exists outside the radiation port or clear progression exists within the radiation port
* Tissue accessible for immunohistochemical evidence of epidermal growth factor receptor expression from a metastatic site (phase II only)
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No unstable angina pectoris
* No symptomatic congestive heart failure
* No cardiac arrhythmia
* No uncontrolled hypertension (systolic blood pressure greater than 150 mm Hg)

Opthalmic

* No abnormalities of the cornea (e.g., severe dry eye syndrome or Sjogren's syndrome)
* No congenital abnormality (e.g., Fuch's dystrophy)
* No abnormal slit-lamp examination using vital dye (e.g., fluorescein or Bengal-Rose)
* No abnormal corneal sensitivity test (e.g., Schirmer test or similar tear-production test)
* Mild dry eye syndrome allowed if patient can use artificial tears and ophthalmologist concurs

Gastrointestinal

* No gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
* No active peptic ulcer disease

Other

* Must be able and willing to undergo a mediport insertion
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except previously excised and inactive basal cell or squamous cell skin cancer
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to erlotinib or other study drugs (e.g., epidermal growth factor inhibitors like cetuximab)
* No significant traumatic injury within the past 3 weeks
* No peripheral neuropathy grade 2 or greater
* No ongoing or active infection
* No other uncontrolled concurrent illness that would preclude study entry
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Phase I:

  * Prior chemotherapy allowed
* Phase II:

  * No prior chemotherapy for metastatic disease
  * Prior adjuvant therapy allowed if disease progresses during adjuvant therapy
  * No prior oxaliplatin

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy and recovered

Surgery

* See Disease Characteristics
* More than 3 weeks since prior major surgery and recovered
* No prior surgical procedures affecting absorption

Other

* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies (commercial or investigational)
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B. Saltz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States